CLINICAL TRIAL: NCT05978648
Title: A Prospective, Multi-cohort, Exploratory Phase II Study of Trilaciclib Combined With Standard Chemotherapy in The Adjuvant Treatment of Hormone Receptor (HR) Negative Breast Cancer
Brief Title: Trilaciclib in Patients With Early-Stage HR-negative Breast Cancer Receiving Adjuvant Chemotherapy
Acronym: SMA-BC-002
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: wang shusen (Other)
Responsible Party: Sponsor-Investigator, wang shusen, Director of Breast Disease Department, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-BC-002
Record Dates: First submitted 2023-07-18; First posted 2023-08-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms
Keywords: Trilaciclib; HR-Negative Breast Cancer; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — trilaciclib; Epirubicin; Cyclophosphamide; Paclitaxel; Docetaxel; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: Triple-negative Breast Cancer (Experimental): Cohort A Administered Trilaciclib in Combination with Chemotherapy(EC-wP)
  Interventions: Drug: Trilaciclib; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- Cohort B: ER-negative PR-negative Her2-positive Breast Cancer (Experimental): Cohort B Administered Trilaciclib in Combination with Chemotherapy(TCbH±P)
  Interventions: Drug: Trilaciclib; Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Trilaciclib — 240 mg/m2, intravenous drip over 30 min within 4 hours before chemotherapy administration on the same day
  Other Names: COSELA®; G1T28
Drug: Epirubicin — 90 mg/m2, intravenous drip, d1, Q3W, 4 cycles.
  Arms: Cohort A: Triple-negative Breast Cancer
Drug: Cyclophosphamide — 600 mg/m2, intravenous drip, d1, Q3W, 4 cycles.
  Arms: Cohort A: Triple-negative Breast Cancer
Drug: Paclitaxel — 80 mg/m2, intravenous drip, d1,8,15, Q3W, 4 cycles.
  Arms: Cohort A: Triple-negative Breast Cancer
Drug: Docetaxel — 75 mg/m2, intravenous drip, d1, Q3W, 6 cycles.
  Arms: Cohort B: ER-negative PR-negative Her2-positive Breast Cancer
Drug: Carboplatin — area under curve(AUC) = 6, intravenous drip, d1, Q3W, 6 cycles.
  Arms: Cohort B: ER-negative PR-negative Her2-positive Breast Cancer
Drug: Trastuzumab — 8 mg/kg in Cycle 1, 6 mg/kg in subsequent cycles, intravenous drip, d1, Q3W, for 1 year.
  Arms: Cohort B: ER-negative PR-negative Her2-positive Breast Cancer
Drug: Pertuzumab — 840mg in Cycle 1, 420mg in subsequent cycles, intravenous drip, d1, Q3W, for 1 year.
  Arms: Cohort B: ER-negative PR-negative Her2-positive Breast Cancer

SUMMARY:
The goal of this multicenter, two-cohort, exploratory clinical trial is to evaluate patients with early stage hormone receptor-negative breast cancer receiving standard adjuvant chemotherapy after surgery. The main question it aims to answer is:

• The efficacy and safety of trilaciclib administered before standard adjuvant chemotherapy regimen using the incidence of grade 3/4 neutropenia as the primary efficacy endpoint.

Participants will divide into two treatment cohorts according to molecular typing type:

* Cohort A will be planned to include post-operative triple-negative breast cancer(TNBC) patients with lymph node positive or tumor > 2 cm treated with trilaciclib combined with epirubicin and cyclophosphamide followed by weekly paclitaxel;
* Cohort B will be planned to include HER2-positive/HR-negative breast cancer patients with axillary node positive or tumor > 2 cm treated with trilaciclib combined with docetaxel, carboplatin and trastuzumab with or without pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* breast cancer meets the following criteria:

  * Histologically or cytologically confirmed and adequately resected non-metastatic primary invasive breast cancer;
  * Cohort A only: ER, PR negative (< 1% nuclear staining as assessed by immunohistochemistry [IHC]), HER2 negative (HER2/CEP17 ratio < 2.0 or mean HER2 gene copy number < 4 signals/nucleus detected by IHC 0 or 1 + or in situ hybridization [ISH]); patients with concurrent bilateral invasive disease met the inclusion criteria if both lesions were HR negative/HER2 negative.
  * Cohort B only: ER, PR negative (< 1% nuclear staining as assessed by immunohistochemistry [IHC]); HER2 positive: HER2/CEP17 ratio ≥ 2.0 or HER2 gene copy number ≥ 4 signals/nucleus detected by IHC 3 + and ISH; HER2 gene copy number ≥ 6 signals/nucleus detected by IHC 3 + or 2 + and ISH); patients with concurrent bilateral invasive disease met the inclusion criteria if both lesions were HR negative/HER2 positive.
  * Subjects must have positive lymph nodes or tumors > 2 cm;
  * The interval between radical surgery and the first dose ≤ 60 days;
* Eastern Cooperative Oncology Group (ECOG) performance score 0-1;
* have appropriate organ function, meet the following criteria: (1) have appropriate bone marrow function: Hb ≥ 100 g/L (no ESA and blood transfusion within 14 days before the first dose); absolute neutrophil count (ANC) ≥ 2 × 10^9/L (no G-CSF within 14 days before the first dose); platelet count ≥ 100 × 10^9/L (no rhTPO/rhIL-11 and platelet transfusion within 14 days before the first dose); (2) appropriate liver and kidney function: alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin (TBIL) ≤ 1.5 × ULN, serum creatinine ≤ 1.5 × ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula); (3) appropriate cardiac function: left ventricular ejection fraction (LVEF) ≥ 55%;
* Non-hematologic toxicities from prior surgical procedures recovered to ≤ Grade 1 or baseline (except alopecia);
* Females of childbearing potential agree to practice reliable contraception during the clinical trial and have a negative serum or urine pregnancy test within 7 days prior to dosing;
* Voluntarily join this study and sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

* Prior neoadjuvant therapy (including chemotherapy, targeted therapy, immunotherapy, or radiotherapy);
* History of other malignancy within 5 years prior to first dose, except basal cell carcinoma and cervical carcinoma in situ;
* Any T4 or N2 or known N3 or M1 breast cancer;
* Subjects who cannot receive or tolerate postoperative chemotherapy for various reasons;
* Heart disease ineligible for epirubicin, docetaxel, trastuzumab/pertuzumab:

  * Any documented history of myocardial infarction, congestive heart failure
  * Angina pectoris requiring antianginal medication
  * Grade 3 or 4 cardiac arrhythmia (NCI CTCAEv5.0)
  * Clinically significant valvular heart disease;
  * Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
* Known history of hypersensitivity to the drug components of this protocol;
* Any other condition that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3/4 neutropenia | Up to 24 weeks
  Proportion of subjects with at least one absolute neutrophil count (ANC) < 1.0 × 10^9/L enrolled and treated with at least one dose of trilaciclib

SECONDARY OUTCOMES:
Neutrophil-related myeloprotective effects | Up to 24 weeks
  Occurrence of febrile neutropenia adverse events(AEs) , and occurrence of Granulocyte colony-stimulating factor(G-CSF) administration
Red blood cell(RBC) -related myeloprotective effects | Up to 24 weeks
  Occurrence of Grade 3/4 decrease of hemoglobin, occurrence and number of RBC transfusions on/after Week 5, and occurrence of erythropoiesis-stimulating agent(ESA) administration
Platelet-related myeloprotective effects | Up to 24 weeks
  Occurrence of Grade 3/4 decrease of platelets, occurrence and number of platelet transfusions, and occurrence of rhTPO/Recombinant human interleukin-11(rhIL-11) administration
Myeloprotective Effects | Up to 24 months
  Hospitalization due to chemotherapy-induced myelosuppression, dose reductions and delays, relative dose intensity(RDI) of chemotherapeutic agents
Safety and tolerability | Up to 24 months
  Incidence of Treatment-Emergent Adverse Events as per CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun-yat sen university cancer center, Guangzhou, Gangdong, China